CLINICAL TRIAL: NCT01047033
Title: Evaluation of Impacts of Health Education for Children of Microcredit Clients in Peru
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Innovations for Poverty Action (Other)
Collaborators: American Medical Women's Association (Other); University of California, Berkeley (Other); Center for Latin American Studies at UCB (Unknown); University of California, San Francisco (Other); Interdisciplinary MPH Program at the UCB School of Public Health (Unknown); Rainer Fund (Unknown)
Responsible Party: Rita Hamad, University of California San Francisco
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: IPA-2007-PE
Record Dates: First submitted 2010-01-08; First posted 2010-01-12 (Estimated); Last update posted 2010-01-12 (Estimated); Status verified 2010-01

CONDITIONS: Child Health Status
Keywords: Poverty; Global health; International health; Latin America; Peru; Child health; Microcredit; Microenterprise; Microfinance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Microcredit only (Active Comparator)
  Interventions: Other: Microcredit
- Microcredit plus health education (Experimental): Thirty minutes of a health education module administered to clients by loan officer at their monthly group meetings over the course of 8 months.
  Interventions: Behavioral: Health education; Other: Microcredit

INTERVENTIONS:
Behavioral: Health education — 30 minutes of a health education module delivered to clients by loan officers during monthly repayment meetings, over the course of 8 months.
  Arms: Microcredit plus health education
Other: Microcredit — Small loans administered to clients through the collaborating microcredit organization, to be repaid monthly over the course of six months in the context of monthly loan group meetings.

SUMMARY:
This purpose of this study is to determine whether a health education intervention for clients of a microcredit organization in Peru will improve health outcomes among clients and their children.

DETAILED DESCRIPTION:
An increasingly popular scheme for poverty alleviation is microcredit, the awarding of small loans to individuals too poor or too remote to take advantage of traditional lending services. Studies have repeatedly shown that income is one of the factors strongly associated with physical and mental wellbeing. Yet economic growth alone doesn't necessarily lead to healthier families, especially if basic health knowledge or health services are absent in the community. Microcredit institutions have recently tried to address this issue by supplementing banking-only microcredit programs with programs that include "tie-ins" or "add-ons" such as health education or health services. A rigorous evaluation of such "banking-plus" endeavors has not yet been conducted, leaving a gap in the knowledge base regarding whether these organizations are meeting their stated goals in catering to both economic and social needs. This study attempts to address this research question using a randomized controlled trial of a health education intervention to clients of a microcredit organization in Peru.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be current clients of the collaborating microcredit organization
* Clients must be at least 18 years of age
* Children of clients must be less than 5 years of age
* Study participants must be able to speak and understand Spanish

Exclusion Criteria:

* Only one client from any particular household may participate

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 2453 (Actual)
Dates: Start 2007-01; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Anthropometric measures including height, weight, and blood hemoglobin level | One year after intervention begins
Client health knowledge on a variety of issues related to child health (e.g. diarrhea, fever) | One year after intervention begins
Child health status as measured by a variety of indicators (e.g. days of diarrhea, presence of bloody diarrhea, presence of severe cough, days of fever, etc.) | One year after intervention begins

SECONDARY OUTCOMES:
Social support as measured by the Duke-UNC FSSQ | One year after intervention begins

CONTACTS AND LOCATIONS:
Overall Officials: Lia Fernald, PhD MBA, Principal Investigator — University of California, Berkeley; Dean Karlan, PhD MBA MPP, Principal Investigator — Yale University
Locations (1):
- Innovations for Poverty Action, Pucallpa, Peru

REFERENCES:
- [Derived] Hamad R, Fernald LCh, Karlan DS. Health education for microcredit clients in Peru: a randomized controlled trial. BMC Public Health. 2011 Jan 24;11(1):51. doi: 10.1186/1471-2458-11-51. PMID 21261988